CLINICAL TRIAL: NCT04585516
Title: Diagnostic Usefulness of Different Types of Gastrointestinal Endoscopic Investigations.
Status: Active, not recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Michiel van Nieuwenhoven, Md, MSc, associate professor, Region Örebro County
Other Study IDs: 274964
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Colo-rectal Cancer; Gastrointestinal Disease
Keywords: colonoscopy; gastroscopy
MeSH Terms: conditions — Colonic Neoplasms; Gastrointestinal Diseases | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patient with suspected colorectal cancer: All patients that were admitted to the department of surgery with suspected colorectal cancer between January 2016 and December 2018 (n=459).
  Interventions: Procedure: endoscopy
- Patients admitted according to the standardized course of care for colorectal cancer: All patients that were admitted to the endoscopy department according to the standardized course of care for colorectal cancer between September 2016 and December 2018 (n=1271).
  Interventions: Procedure: endoscopy
- Patients < 50 years that were admitted for gastroscopy: All patients younger than 50 years that were admitted to the endoscopy department for a gastroscopy between jan 2018 and April 2019 (n= 1915)
  Interventions: Procedure: endoscopy
- Patients >80 years that were admitted for colonoscopy: All patients older than 80 years that were admitted to the endoscopy department for a colonoscopy between Sept 2016 and Jan 2019 (n= 981)
  Interventions: Procedure: endoscopy

INTERVENTIONS:
Procedure: endoscopy — Colonoscopy or gastroscopy

SUMMARY:
The number of endoscopies performed varies greatly between different countries and does not reflect variations in disease incidents. The costs of unnecessary endoscopies are significant and with a better selection of which patients need to be examined with endoscopy, resources could be saved in healthcare, and a better triage would mean that malignancies and other more serious conditions do not have to wait. An example of unnecessary endoscopy is a colonoscopy in patients with irritable bowel syndrome or gastroscopy in patients with functional dyspepsia.

The purpose of the project is, among other things:

* What diagnostic benefit have gastroscopy, colonoscopy, capsule endoscopy and double balloon enteroscopy for different indications in different age groups?
* What are the risks of this type of examination?
* Can patients be better selected based on symptoms, psychometric data or laboratory findings to reduce the number of unnecessary examinations and prioritize those that should be scooped up first?
* Can changed calling methods reduce the number of late cancellations and rebookings and missed patients?

DETAILED DESCRIPTION:
1: Identification of colorectal cancer in Örebro Region - Effectiveness of Standardised Course of Care.

Introduction: To shorten time to diagnosis of suspected colorectal cancer (CRC) in Sweden, CRC was included in the "standardised course of care" (SCC) in 2016. However, not all patients with CRC are referred via the SCC, and CRC is also found in patients undergoing a routine colonoscopy.

Objective: To identify CRC cases in the Örebro Region and how they were identified. Furthermore, to investigate the reasons for and possible effect of not being included in the SCC-CRC for cases found via colonoscopy.

Methods: Reviewing medical records of patients with CRC referred to the Clinic of Surgery in the Örebro Region in 2016-2018 (n=459).

The information recalled from the journals includes diagnostic pathway of CRC discovery, age, gender, Body Mass Index (BMI), Hb-value, date of referral to colonoscopy, date of preformed colonoscopy, referral route (SCC-CRC or non-CRC-SCC), reasons for referral (including SCC-CRC criteria) and patient symptoms. Furthermore, we will gather data of tumor localization (caecum; ascending colon; splenic flexure; transverse colon; hepatic flexure; descending colon; sigmoid and rectum), TNM-stage of the tumor, [11] tumor differentiation (high grade or low grade tumor), and source of referral (referral by general practitioner or referral by hospital physician).

Age is determined at the time of referral. BMI is defined as the most recent BMI value at time of referral within six months prior or six months after referral date. Hb-value will be defined as the most recent Hb-value within a month prior of the time of referral. Diagnostic interval is defined as the number of days days between the referral and the colonoscopy. When the tumor localization is described as in between two locations of the colon (e.g. descendent colon and sigmoid colon) the most proximal location is chosen for statistical analysis. Patients with two or more synchronous cancers are registered as more than one incident per case. When the tumor localization is described as being present in the rectosigmoid transition, the sigmoid is used as the tumor localization in the analysis. When patients have two or more symptoms and reasons for referral, data are registered as more than one incident per case. TNM stage is converted to tumor stage I-IV. [1] When patients have one or more synchronic cancer with different TNM stages, the highest cancer stage is chosen for analysis. If the TNM stage is not fully known (e.g. information about lymph nodes and metastases are missing) the stage is set as no lymph node engagement or metastases, If the original referral cannot be found, date and reasons for referral are collected from journal entries.

2: The Swedish standardized course of care for colorectal cancer - cancer prevalence and predictive values of entry criteria.

Introduction: To shorten waiting times for cancer treatment and to reduce national inequalities in cancer care, the standardized course of care (SCC) was implemented in Sweden. The SCC for colorectal cancer (CRC-SCC) was implemented in 2016. Since then, about 46.000 patients have been examined according to a CRC-SCC. However, few studies have been conducted to evaluate the CRC-SCC.

Aim: To identify the prevalence of colorectal cancer (CRC) in patients referred to Örebro University Hospital (USÖ) according to a CRC-SCC. We also aimed to investigate the positive predicting values (PPVs) and odds ratios (ORs) of different SCC-criteria with respect to CRC.

Method: Medical record review including all patients examined by colonoscopy as part of a CRC-SCC-referral to USÖ between September, 2016 and December 2018 (n=1271).The parameters of interest include; patient characteristics such as sex and age, the SCC-criteria for reasonable suspicion of cancer. If the patient has an altered bowel function it is registered whether the patient has loose stool, constipation, a combination of the two, or not specified in the referral. Rectal bleeding is defined as fresh rectal bleeding, excluding melaena. Patients who fulfill multiple criteria are registered as more than one incidence case. Laboratory values such as fecal occult blood, plasma-hemoglobin, and fecal-calprotectin (F-calprotectin) are registered. The most resent value at the time of referral is used. If there is no value within a month of the referral, no value was registered. A patient is regarded to have a positive fecal occult blood test (FOBT) if at least one out of three tests is positive. A f-calprotectin <50mg/kg is considered negative. Findings from the colonoscopy such as CRC, polyps, inflammation of the colon, diverticulosis, hemorrhoids, angiodysplasia or no finding are registered. All findings with colonoscopy are, if possible, histologically verified.

3: Why do we perform gastroscopy in younger patients?

Background: Esophagogastroduodenoscopy (EGD) is the golden standard diagnostic method in upper GI pathologies. The current guidelines indicate that patients with alarm symptoms and/or dyspeptic patients over 50 years of age should be readily investigated with gastroscopy. However, EGD is also frequently performed in the younger population, where it often results in absence of pathological findings. In Örebro approximately 4000 EGD are completed yearly, approximately 40% of the EGD's are performed in patients >50 years, requiring extensive resources.

Aim: to identify factors in the EGD referrals of patients under 50 years of age without alarm symptoms, in order to minimize the number of unnecessary EGD's in this age group.

Method and material: The study will be conducted as a retrospective database study. We will process the EGD referrals and diagnostic findings of young patients (age 18-50 y) performed during 2017-2019 at Örebro University Hospital. Statistical analysis will be performed to identify which signs and symptoms are associated with a pathological finding during EGD and which signs and symptoms are associated with a negative finding. The parameters of interest include; patient characteristics such as sex and age will separately analyze the groups 18-29y, 30-39y, and 40-49 y. Other parameters include: BMI, ethnicity, use of NSAID/ASA, h. pylori analysis, eventual treatment for h. pylori, smoking, alcohol consumption,presence of GI disease before gastroscopy, previously done gastroscopy, source of referral (primary health care or in-hospital patients), if present: fulfillment of Rome IV criteria for functional dyspepsia, symptoms such as anemia, fecal occult blood, palpable mass in abdomen, weight loss, loss of appetite, dysphagia, vomiting, jaundice, waiting time between referral and gastroscopy, as well as the findings under gastroscopy; GERD/oesofagitis, peptic ulcus, gastritis, dysplasia/cancer, IBD, celiac disease, hiatal hernia

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent a diagnostic diagnostic procedure at the endoscopy unit at the University Hospital Örebro.

Exclusion Criteria:

Patients <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent an endoscopic diagnostic procedure.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
All confirmed colorectal cancer cases that were diagnosed via colonoscopy. | between September 2016 and December 2018
  The proportion of patients that was admitted to the department of surgery with confirmed colorectal cancer, diagnosed according to the standardized course of care for colorectal cancer.
Proportion of patients that was diagnosed with colorectal cancer. with colorectal cancer | between September 2016 and December 2018
  All patients that were admitted to the endoscopy unit according to the standardized course of care for colorectal cancer.
Presence of upper GI pathology | between Jan 2019-April 2020
  The proportion of upper GI pathology in all patients <50 years who were admitted for a gastroscopy

SECONDARY OUTCOMES:
route of colorectal cancer diagnosis 1 | January 2016 and December 2018
  The proportion of patients with confirmed colorectal cancer that was diagnosed with colonoscopy according to the standardized chain of care for colorectal cancer.
route of colorectal cancer diagnosis 2 | January 2016 and December 2018
  The proportion of patients with confirmed colorectal cancer that was diagnosed with routine colonoscopy.
Localization of colorectal cancer | January 2016 and December 2018
  The site of the tumor in confirmed colorectal cancer
tumor characteristics of colorectal cancer 1 | January 2016 and December 2018
  The stage of the tumor in confirmed colorectal cancer
tumor characteristics of colorectal cancer 2 | January 2016 and December 2018
  The histology of the tumor in confirmed colorectal cancer
symptom characteristics of colorectal cancer 1 | January 2016 and December 2018
  proportion of patients with changes in bowel habits >4 weeks in patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 2 | January 2016 and December 2018
  proportion of patients with radiology in patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 3 | January 2016 and December 2018
  proportion of patients with abnormal rectal finding via palpation or rectoscopy in patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 4 | January 2016 and December 2018
  proportion of patients with rectal bleeding without obvious source in patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 5 | January 2016 and December 2018
  proportion of patients with rectal bleeding despite adequate treatment of bleeding source in patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 6 | January 2016 and December 2018
  proportion of patients with rectal bleeding in high-risk patients with confirmed colorectal cancer
symptom characteristics of colorectal cancer 7 | January 2016 and December 2018
  proportion of patients with bleeding anemia of unknown source in patients with confirmed colorectal cancer
patient characteristics of colorectal cancer 1 | January 2016 and December 2018
  male/female
patient characteristics of colorectal cancer 2 | January 2016 and December 2018
  age
patient characteristics of colorectal cancer 3 | January 2016 and December 2018
  hemoglobine value
patient characteristics of colorectal cancer 4 | January 2016 and December 2018
  calprotectin value
patient characteristics of colorectal cancer 5 | January 2016 and December 2018
  Days between referral and colonoscopy
patient characteristics of colorectal cancer 6 | January 2016 and December 2018
  referral from primary health care yes/no
patient characteristics of colorectal cancer 7 | January 2016 - December 2018
  referral year: 2017/2017/2018

OTHER OUTCOMES:
Patient characteristics in patients who were admitted for colonoscopy 1 | September 2016 - December 2018
  proportion of patients with weight loss >10%
Patient characteristics in patients who were admitted for colonoscopy 2 | September 2016 - December 2018
  age
Patient characteristics in patients who were admitted for colonoscopy 3 | September 2016 - December 2018 0
  male/female
symptom characteristics in patients who were admitted for colonoscopy 1 | September 2016 - December 2018
  proportion of patients with loose stools
symptom characteristics in patients who were admitted for colonoscopy 2 | September 2016 - December 2018
  proportion of patients with constipation
symptom characteristics in patients who were admitted for colonoscopy 3 | September 2016 - December 2018
  proportion of patients with altered bowel function specified
symptom characteristics in patients who were admitted for colonoscopy 4 | September 2016 - December 2018
  proportion of patients with abnormal radiology
symptom characteristics in patients who were admitted for colonoscopy 5 | September 2016 - December 2018
  proportion of patients with abnormal rectal examination
symptom characteristics in patients who were admitted for colonoscopy 6 | September 2016 - December 2018
  proportion of patients with rectal bleeding without obvious source
symptom characteristics in patients who were admitted for colonoscopy 7 | September 2016 - December 2018
  proportion of patients with rectal bleeding despite adequate treatment
symptom characteristics in patients who were admitted for colonoscopy 8 | September 2016 - December 2018
  proportion of high-risk patients with rectal bleeding
symptom characteristics in patients who were admitted for colonoscopy 9 | September 2016 - December 2018
  proportion of patients with anemia of unknown cause
symptom characteristics in patients who were admitted for colonoscopy 10 | September 2016 - December 2018
  proportion of patients with positive fecal occult blood test
symptom characteristics in patients who were admitted for colonoscopy 11 | September 2016 - December 2018
  proportion of patients with increased fecal calprotectin
Endoscopic finding in patients who were admitted for colonoscopy 1 | September 2016 - December 2018
  Proportion of patients with polyps high-grade/low grade dysplasia
Endoscopic finding in patients who were admitted for colonoscopy 2 | September 2016 - December 2018
  Proportion of patients with diverticulosis
Endoscopic finding in patients who were admitted for colonoscopy 3 | September 2016 - December 2018
  Proportion of patients with inflammation unspecified
Endoscopic finding in patients who were admitted for colonoscopy 4 | September 2016 - December 2018
  Proportion of patients with IBD
Endoscopic finding in patients who were admitted for colonoscopy 5 | September 2016 - December 2018
  Proportion of patients with infectious colitis
Endoscopic finding in patients who were admitted for colonoscopy 6 | September 2016 - December 2018
  Proportion of patients with microscopic colitis
Endoscopic finding in patients who were admitted for colonoscopy 7 | September 2016 - December 2018
  Proportion of patients with diverticulitis
Endoscopic finding in patients who were admitted for colonoscopy 8 | September 2016 - December 2018
  Proportion of patients with hemorrhoids
Endoscopic finding in patients who were admitted for colonoscopy 9 | September 2016 - December 2018
  Proportion of patients with angiodysplasia
Endoscopic finding in patients who were admitted for colonoscopy 10 | September 2016 - December 2018
  Proportion of patients with no findings.
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 1 | Jan 2019-April 2020
  proportion of patients with weight loss >10%
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 2 | Jan 2019-April 2020
  proportion of patients with loss of appetite
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 3 | Jan 2019-April 2020
  proportion of patients with dysphagia
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 4 | Jan 2019-April 2020
  proportion of patients with vomiting
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 5 | Jan 2019-April 2020
  proportion of patients with jaundice
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 6 | Jan 2019-April 2020
  proportion of patients with GERD/oesofagitis
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 7 | Jan 2019-April 2020
  proportion of patients with gastritis
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 8 | Jan 2019-April 2020
  proportion of patients with peptic ulcer disease
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 9 | Jan 2019-April 2020
  proportion of patients with dysplasia/cancer
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 10 | Jan 2019-April 2020
  proportion of patients with IBD
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 11 | Jan 2019-April 2020
  proportion of patients with celiac disease
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 12 | Jan 2019-April 2020
  proportion of patients who meet Rome IV criteria for functional dyspepsia.
Symptom characteristics in patients < 50 years who were admitted for a gastroscopy 13 | Jan 2019-April 2020
  proportion of patients with other unspecified pathology
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 1 | Jan 2019-April 2020
  male/female
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 2 | Jan 2019-April 2020
  proportion of patients who smoke
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 3 | Jan 2019-April 2020
  proportion of patients with age 18-29, age 30-39, age 40-49.
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 4 | Jan 2019-April 2020
  proportion of patients using NSAIDs/ASA
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 5 | Jan 2019-April 2020
  proportion of patients who had done a h. pylori test
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 6 | Jan 2019-April 2020
  proportion of patients with a positive h. pylori test
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 7 | Jan 2019-April 2020
  proportion of patients who were eradicated after a positive h. pylori test
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 8 | Jan 2019-April 2020
  ethnicity of patients (proportion caucasian origin, African origin, arabic origin, asian origin)
Patients characteristics in patients < 50 years who were admitted for a gastroscopy 9 | Jan 2019-April 2020
  days between referral and gastroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Örebro, Egion Rebro Ounty, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen L, Rasanen N, Berggren F, van Nieuwenhoven MA. Assessing age-related risks of gastrointestinal pathologies: a comparative study of gastroscopy outcomes across decades. Therap Adv Gastroenterol. 2024 Oct 28;17:17562848241290446. doi: 10.1177/17562848241290446. eCollection 2024. PMID 39474441
- [Derived] Andersson E, Nyhlin N, van Nieuwenhoven MA. The effectiveness of the colorectal cancer referral pathway - identification of colorectal cancer in a Swedish region. Scand J Gastroenterol. 2021 May;56(5):552-558. doi: 10.1080/00365521.2021.1899276. Epub 2021 Mar 22. PMID 33749502